CLINICAL TRIAL: NCT03034499
Title: Single Versus Multi-port Robotic Assisted Sacrocolpopexy for Repair of Vaginal Apex Prolapse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, ROY LAUTERBACH MD, Principal investigator, Rambam Health Care Campus
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0631-16-RMB
Record Dates: First submitted 2017-01-25; First posted 2017-01-27 (Estimated); Last update posted 2019-06-11 (Actual); Status verified 2019-06

CONDITIONS: Pelvic Organ Prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single-port sacrocolpopexy (Active Comparator): Patients with vaginal apex prolapse randomized to undergo repair by single-port sacrocolpopexy.
  Interventions: Procedure: Single-port sacrocolpopexy
- Multi-port sacrocolpopexy (Active Comparator): Patients with vaginal apex prolapse randomized to undergo repair by multi- port sacrocolpopexy.
  Interventions: Procedure: Multi-port sacrocolpopexy

INTERVENTIONS:
Procedure: Single-port sacrocolpopexy — Single-port sacrocolpopexy surgery for the repair of vaginal apex prolapse.
  Arms: Single-port sacrocolpopexy
Procedure: Multi-port sacrocolpopexy — Multi-port sacrocolpopexy surgery for the repair of vaginal apex prolapse.
  Arms: Multi-port sacrocolpopexy

SUMMARY:
A prospective randomized controlled study intended to compare the efficacy of 2 methods of robotic assisted sacrocolpopexy for the repair of vaginal apex prolapse:

1. Via single-port.
2. Via multi-port.

DETAILED DESCRIPTION:
One hundred female patients diagnosed with vaginal apex prolapse will be recruited to a prospective randomized controlled study intended to compare the efficacy of 2 methods of robotic assisted sacrocolpopexy:

1. Via single-port.
2. Via multi-port. The patients will be evaluated and randomized 2 weeks before the expected date of surgery during which eligibility will be examined.

Patients' electronic files will be reviewed post operatively to acquire information regarding medical history, prolapse scores, surgical information, anesthesia information and surgical complications.

Patients will have 3 week and 3 month post operative follow-up sessions to determine surgical success, late complications and patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Female patients with vaginal apex prolapse that are eligible for repair by sacrocolpopexy.

Exclusion Criteria:

* Patients after previous hysterectomy.
* Patients after previous surgical procedures for prolapse repair.

Ages: 30 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female patients.
Enrollment: 80 (Actual)
Dates: Start 2017-03-20 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
Comparison of surgical time | Up to four months (2 weeks before surgery until 3 months post-surgery).
  Comparison of surgical time in single versus multi-port robotic assisted sacrocolpopexy.

SECONDARY OUTCOMES:
Comparison of surgical success | Up to four months (2 weeks before surgery until 3 months post-surgery).
  Comparison of surgical success in single versus multi-port robotic assisted sacrocolpopexy.
Comparison of surgical complications | Up to four months (2 weeks before surgery until 3 months post-surgery).
  Comparison of surgical complications (including bleeding and post operative pain) in single versus multi-port robotic assisted sacrocolpopexy.

CONTACTS AND LOCATIONS:
Overall Officials: Roy Lauterbach, MD, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam health care campus, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Matanes E, Boulus S, Lauterbach R, Amit A, Weiner Z, Lowenstein L. Robotic laparoendoscopic single-site compared with robotic multi-port sacrocolpopexy for apical compartment prolapse. Am J Obstet Gynecol. 2020 Apr;222(4):358.e1-358.e11. doi: 10.1016/j.ajog.2019.09.048. Epub 2019 Oct 4. PMID 31589864